CLINICAL TRIAL: NCT03480958
Title: Comparison of Erector Spinae Plane Block With Thoracic Paravertebral Block for Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Yavuz Gurkan, Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-94
Record Dates: First submitted 2018-03-18; First posted 2018-03-29 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Postoperative Pain; Breast Cancer
Keywords: erector spinae plane block; thoracic paravertebral block; breast surgery; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESP group (Active Comparator): Erector Spinae Plane Block administered group
  Interventions: Device: Intravenous morphine patient controlled device; Other: Erector Spinae Plane Block
- TPVB group (Active Comparator): Thoracic Paravertebral Block administered group
  Interventions: Device: Intravenous morphine patient controlled device; Other: Thoracic Paravertebral Block
- Control Group (Other): No regional anesthesia technique will be applied to control group; but will be provided with iv PCA
  Interventions: Device: Intravenous morphine patient controlled device

INTERVENTIONS:
Device: Intravenous morphine patient controlled device — 24 hour morphine consumption will be recorded
Other: Erector Spinae Plane Block — erector spinae plane block will be administered before the surgery
  Arms: ESP group
Other: Thoracic Paravertebral Block — thoracic paravertebral block will be administered before the surgery
  Arms: TPVB group

SUMMARY:
Postoperative analgesia in breast surgery is a difficult and overworked issue due to etensive surgery and complex innervation of the breast. Erector spinae plane block (ESB) is a new defined and promising regional anesthesia technique for thoracic analgesia. Main purpose of this study is to compare the analgesic effect of ultrasound guided ESB with thoracic paravertebral block - the golden standard method for postoperative regional analgesia technique in breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* 25-70 years of agge
* ASA I-II
* Undergoing elective breast cancer surgery

Exclusion Criteria:

* obesity (body mass index >35 kg/m2)
* infection of the skin at the site of needle puncture area
* patients with known allergies to any of the study drugs
* coagulopathy
* recent use of analgesic drugs

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 24 hour postoperatively
  All patients will be provided with IV morphine PCA and morphine consumption after 24 hour postoperatively will be recorded.

SECONDARY OUTCOMES:
Numering Rating Scale scores for pain | 24 hour
  Numeric Rating Scale (NRS) for pain will be used. The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain. It is for adults and children 10 years old or older. 0 means no pain and 10 means most imaginable pain
Postoperative nausea and vomiting | 24h
  Incidence of postoperative nausea and vomiting will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gurkan Y, Aksu C, Kus A, Yorukoglu UH. Erector spinae plane block and thoracic paravertebral block for breast surgery compared to IV-morphine: A randomized controlled trial. J Clin Anesth. 2020 Feb;59:84-88. doi: 10.1016/j.jclinane.2019.06.036. Epub 2019 Jul 4. PMID 31280100